CLINICAL TRIAL: NCT02719145
Title: Circulating Micro RNAs Expression in Egyptian Bronchial Asthma and COPD Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Adel Salah Bediwy, Professor, Tanta University
Other Study IDs: TFMEC1015
Record Dates: First submitted 2016-03-19; First posted 2016-03-25 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Asthma; COPD
Keywords: micro RNA; asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control group (group 1): 10 healthy volunteer subjects.
- Asthma group (group 2): 10 asthmatic patients.
- COPD group (group 3): 10 COPD patients.

SUMMARY:
This cross sectional study will be carried out on 30 subjects who will be recruited from the outpatient clinic of Chest Department, Tanta University Hospital.

They will be classified into 3 groups:

Group I: It will include 10 healthy volunteer subjects. Group II: It will include 10 asthmatic patients. Group III: It will include 10 COPD patients. miR-7, miR-20a, miR-21, miR-22, miR-145 and miR-155 will be measured in serum samples from all subjects

DETAILED DESCRIPTION:
The following will be done for all subjects:

1. Thorough history taking with stress on age, age at onset, duration of the disease, smoking history, therapeutic history with stress on their drugs, course of the disease, history of any previous attacks of acute severe asthma or exacerbation of COPD.
2. Complete physical examination.
3. Chest x-ray P.A view.
4. Complete blood picture.
5. Ventilatory function tests including FVC, FEVI and FEVI/FVC, PEFR and FEF25-75% using computerized spirometry apparatus.

Quantitative assessment of miRNA levels: will be used to assay miR-7, miR-20a, miR-21, miR-22, miR-145 and miR-155 in serum samples from all subjects. These miRNAs were selected based on prediction algorithms that suggested that these miRNAs were involved in the regulation of cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: healthy volunteers with no history of chest troubles.
* Group 2: 10 asthmatic patients with history of paroxysmal wheezing, dyspnea, chest distress, and/or coughing; with Reversible airflow limitation as will be measured by an increase in forced expiratory volume in one second (FEV1) of at least 12% and of more than 200 ml after inhalation of 200 μg salbutamol.
* Group 3: 10 COPD patients who have chronic airﬂow limitation on spirometry (FEV1/FVC is less than 0.7), and the patients have irreversible airflow limitation as will be measured by an increase in (FEV1) by less than12% or less than 200 ml after inhalation of 200 μg salbutamol.

Exclusion Criteria:

* Upper or lower respiratory tract infection during the month preceding the study.
* Other chronic respiratory or systemic illness.
* Usage of systemic steroids within 2 months prior to the study.
* Inability to provide informed consent or who refused to draw off blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross sectional study will be carried out on 30 subjects who will be recruited from the outpatient clinic of Chest Department, Tanta University Hospital.
  They will be classified into 3 groups:
  Group I: It will includ 10 healthy volunteer subjects. Group II: It will include 10 asthmatic patients. Group III: It will include 10 COPD patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
miR-7, miR-20a, miR-21, miR-22, miR-145 and miR-155 in serum samples from control, asthma and COPD Egyptian subjects. | 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Adel S Bediwy, MD, Study Chair — Chest Department, Faculty of Medicine, Tanta University; Salwa A Ganna, MD, Principal Investigator — Chest Department, Faculty of Medicine, Tanta University; Said Hammad, MD, Principal Investigator — Clinical Pathology Department, Faculty of Medicine, Tanta University; Abdel-Aziz A Zidan, PHD, Principal Investigator — Director of Genomics and Proteomics Unit, Center of Excellence in Cancer Research, Tanta University
Locations (1):
- Chest Department, Faculty of Medicine, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Van Pottelberge GR, Mestdagh P, Bracke KR, Thas O, van Durme YM, Joos GF, Vandesompele J, Brusselle GG. MicroRNA expression in induced sputum of smokers and patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2011 Apr 1;183(7):898-906. doi: 10.1164/rccm.201002-0304OC. Epub 2010 Oct 29. PMID 21037022
- [Result] Wang Y, Yang L, Li P, Huang H, Liu T, He H, Lin Z, Jiang Y, Ren N, Wu B, Kamp DW, Tan J, Liu G. Circulating microRNA Signatures Associated with Childhood Asthma. Clin Lab. 2015;61(5-6):467-74. doi: 10.7754/clin.lab.2014.141020. PMID 26118177